CLINICAL TRIAL: NCT03739125
Title: Efficacy and Safety of CKD-501 Added to D150 Plus D745 10mg Therapy in Patients With Type 2 Diabetes Inadequately Controlled With D150 Plus D745 10mg: Multi-center, Randomized, Double-blind, Parallel-group, Placebo Control, Therapeutic Confirmatory Study
Brief Title: Efficacy and Safety of CKD-501 Added to D150 Plus D745 10mg Therapy in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19DM16022
Record Dates: First submitted 2018-02-22; First posted 2018-11-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — lobeglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-501 0.5mg (Experimental): CKD-501 0.5mg
  Interventions: Drug: CKD-501 0.5mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CKD-501 0.5mg — CKD-501 0.5mg, orally, 1 tablet once a day for 24weeks or 52weeks(if extension study) with D150 and D745
  Other Names: Lobeglitazone
  Arms: CKD-501 0.5mg
Drug: Placebo — orally, 1 tablet once a day for 24weeks or 52weeks(if extension study) with D150 and D745
  Arms: Placebo

SUMMARY:
The purpose of this study is to prove that the group treated with CKD-501 in combination added that the reduction of glycated hemoglobin superior to placebo treated group added in combination.

DETAILED DESCRIPTION:
The aim of this phase III study was to evaluate the efficacy and safety of additional combined CKD-501 administration for 24 weeks in patients with type 2 diabetes who were not adequately controlled for blood glucose by the combination of D150 and D745 10mg .

Furthermore, the extension study for additional 28 weeks is designed to confirm long term safety of CKD-501 as an oral hypoglycemic agent.

ELIGIBILITY:
Inclusion Criteria:

* Between 19 years and 75 years old(male or female)
* Type Ⅱ diabetes mellitus
* The patient who has been taking oral hypoglycemic agent at least 8weeks with HbA1c 7 to 10% at screening test
* BMI between 21kg/㎡ and 40kg/㎡
* C-peptide level is over 1.0 ng/ml
* Agreement with written informed consent
* HbA1c 7 to 10% after Run-in period

Exclusion Criteria:

* Type I diabetes or secondary diabetes
* Continuous or non continuous treatment(over 7 days) insulin within 3 months prior to screening
* Treatment with TZD within 3months or patient who have experience such as hypersensitivity reaction, serious adverse event or no effect by treatment with TZD, SGLT2, BU
* Chronic(continuous over 7 days) oral or non oral corticosteroids treatment within 1 month prior to screening
* Treatment with anti-obesity drugs within 3months
* Past history: lactic acidosis or metformin contraindication
* Acute or chronic metabolic acidosis including diabetic ketoacidosis
* History of proliferative diabetic retinopathy
* Severe infection, severe injury patients, patients of pre and post operation
* Patients with urinary tract infection including urinary tract sepsis and pyelonephritis
* Malnutrition, weakness, starvation, hyposthenia, pituitary insufficiency or adrenal insufficiency
* History of malignant tumor within 5years
* Drug abuse or history of alcoholism
* Severe pulmonary dysfunction, severe GI disorder
* History of myocardial infarction, heart failure, cerebral infarction, cerebral hemorrhage or unstable angina within 6 months
* Fasting Plasma Glucose level is over 270 mg/dl
* Triglyceride level is 500 mg/dl and over
* Significant abnormal liver dysfunction
* Anemia
* Abnormality of thyroid function(out of significant normal TSH range )
* eGFR is less than 60ml/min/1.73m^2
* Pregnant women or nursing mothers
* Fertile women who not practice contraception with appropriate methods
* Participated in other trial within 4 weeks
* Participating in other trial at present
* In investigator's judgment

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Glycosylated Hemoglobin (HbA1c) | Baseline, 24 weeks

SECONDARY OUTCOMES:
Change from baseline in Glycosylated Hemoglobin (HbA1c) | Baseline, 52 weeks
Change from baseline in Fasting plasma glucose | Baseline, 24 weeks, 52weeks
Change from baseline in HOMA-IR(Homeostasis Model Assessment of Insulin Resistance) | Baseline, 24 weeks, 52weeks
Change from baseline in HOMA-β(Homeostasis Model Assessment of β-cell function) | Baseline, 24 weeks, 52weeks
Change from baseline in QUICKI(Quantitative Insulin Check Index) | Baseline, 24 weeks, 52weeks
HbA1c target achievement rate at 24, 52weeks(HbA1c < 6.5%, 7%) | Baseline, 24 weeks, 52weeks
Change from baseline in Total Cholesterol | Baseline, 24 weeks, 52weeks
Change from baseline in Triglycerides | Baseline, 24 weeks, 52weeks
Change from baseline in LDL-Cholesterol | Baseline, 24 weeks, 52weeks
Change from baseline in HDL-Cholesterol | Baseline, 24 weeks, 52weeks
Change from baseline in non-HDL-Cholesterol | Baseline, 24 weeks, 52weeks
Change from baseline in Small Dense LDL-Cholesterol | Baseline, 24 weeks, 52weeks
Change from baseline in FFA(Free Fatty Acid) | Baseline, 24 weeks, 52weeks
Change from baseline in Apo-AⅠ | Baseline, 24 weeks, 52weeks
Change from baseline in Apo-B | Baseline, 24 weeks, 52weeks
Change from baseline in Apo-CⅢ | Baseline, 24 weeks, 52weeks
Evaluate safety of CKD-501 from number of participants with adverse events | Baseline, 24 weeks, 52weeks

CONTACTS AND LOCATIONS:
Overall Officials: BongSoo Cha, Ph.D, Study Chair — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No